CLINICAL TRIAL: NCT04864379
Title: Safety, Tolerability and Immunogenicity of a Personalized Neoantigen Cancer Vaccine Combined With Anti-PD-1 and Radiofrequency Ablation in Patients With Advanced Solid Tumors
Brief Title: Clinical Study of a Personalized Neoantigen Cancer Vaccine Combined With Anti-PD-1 and RFA in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yong Fang, Chief Physician, Sir Run Run Shaw Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INEO-P-003
Record Dates: First submitted 2021-04-25; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Advanced Malignant Solid Tumor
MeSH Terms: interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Adjuvants, Immunologic; Colony-Stimulating Factors; Immune Checkpoint Inhibitors; Radiofrequency Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA+PD-1+iNeo-Vac-P01 (Experimental): Patients will undergo radiofrequency ablation. At Week 3, patients will receive PD-1 at a dose of 200mg administered by intravenous infusion (IV) every 2 weeks. At Week 12,all patients,regardless of their disease status,iNeo-Vac-P01(300mcg per peptide)+ GM-CSF (40mcg) on days 1, 4, 8, 15, 22, 52, and 82 from week 12. Additional booster vaccines might be administered depending on ethics and patients' potential benefit.
  Interventions: Biological: iNeo-Vac-P01; Other: GM-CSF; Drug: PD-1; Procedure: RFA
- RFA+iNeo-Vac-P01+PD-1 (Experimental): Patients will undergo radiofrequency ablation. At Week 12, patients will receive iNeo-Vac-P01(300mcg per peptide)+ GM-CSF (40mcg) on days 1, 4, 8, 15, 22, 52, and 82 from week 12. Additional booster vaccines might be administered depending on ethics and patients' potential benefit. At Week 16, patients,regard of their disease status,will receive PD-1 at a dose of 200mg administered by intravenous infusion (IV) every 2 weeks.
  Interventions: Biological: iNeo-Vac-P01; Other: GM-CSF; Drug: PD-1; Procedure: RFA

INTERVENTIONS:
Biological: iNeo-Vac-P01 — iNeo-Vac-P01: 300 mcg per peptide
  Other Names: Neoantigen peptides
Other: GM-CSF — GM-CSF: 40 mcg
  Other Names: immune adjuvant; granulocyte-macrophage colony stimulating factor
Drug: PD-1 — PD-1: 200mg administered by intravenous infusion every 2 weeks.
  Other Names: PD-1 inhibitor
Procedure: RFA — Radiofrequency ablation surgery
  Other Names: Radiofrequency ablation

SUMMARY:
This research study is evaluating a new type of personalized neoantigen cancer vaccine（iNeo-Vac-P01）combined with anti-PD-1 antibody and radiofrequency ablation as a possible treatment for patients with advanced solid tumors. The primary objective of this trial is to evaluate safety, tolerability and immunogenicity of iNeo-Vac-P01 in combination with anti-PD-1 and radiofrequency ablation, so as to provide a new personalized therapeutic strategy for patients.

It is known that cancer patients have mutations (changes in genetic material) that are specific to an individual patient and tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune responses, which may help the participant's body fight any tumor cells that could cause the cancer to come back in the future. The study will examine the safety of the vaccine when given at several different time points and will examine the participant's blood cells for signs that the vaccine induced an immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Must freely sign informed consent;
2. Aged 18 to 75 years old;
3. Life expectancy of greater than 3 months.
4. At least one measurable lesion according to RECIST 1.1 criteria(Radiofrequency ablation of lesions was excluded).
5. histologically confirmed Advanced solid tumors,
6. have failed standard treatment, or unsuitable to receive standard treatment
7. Liver metastases are present and are suitable for radiofrequency ablation；
8. agreeable to allow tumor and normal samples to be submitted for complete exome and transcription sequencing.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
10. Good hematopoietic function ， defined as absolute neutrophils count ≥1.5×109 /L, platelet count ≥100 ×109 /L, and hemoglobin ≥90g/L；
11. Good liver function, defined as total bilirubin levels ≤1.5 times the upper normal limit (ULN), and glutamic-oxalacetic transaminase (AST) and glutamic-pyruvic transaminase (ALT) levels ≤5 times ULN;
12. Good renal function, defined as serum creatinine ≤1.5 times ULN or calculated creatinine clearance ≥ 60 mL /min (Cockcroft-Gault formula); Routine urine examination urine protein less than 2+, or 24 hours urine protein quantitative <1g;
13. Good coagulation function, defined as INR or prothrombin time (PT) ≤1.5 times ULN; If the subject is receiving anticoagulant therapy, PT is acceptable as long as it is within the range of anticoagulant drug use；
14. Pregnant, lactating women and women of child-bearing age must have a negative pregnancy test within 7 days before entering the group, and short-term have no fertility plan, and are willing to take protective measures (contraception or other birth control methods) before and during the clinical trial;

Exclusion Criteria:

1. Currently participating in an interventional clinical study treatment or has received other investigational drugs or used investigational devices within 4 weeks prior to the first administration;
2. Major surgical treatment within 3 weeks prior to first administration;
3. Completed palliative radiotherapy within 7 days prior to first administration;
4. Clinical active diverticulitis, abdominal abscess, and gastrointestinal obstruction;
5. Have none suitable neoantigen;
6. Have been bone marrow or stem cell transplants;
7. Clinically uncontrollable pleural effusion/peritoneal effusion/pericardial effusion;
8. Severe known allergic reactions (≥ grade 3) to the active ingredient and/or any excipient of PD-1 monoclonal antibody；
9. Active autoimmune disease requiring systemic treatment occurred within 2 years prior to initial administration；
10. Diagnosed with immunodeficiency or was receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dosing of the study；
11. Full recovery from toxicity and/or complications associated with any intervention has not been achieved prior to the commencement of treatment；
12. Other tumors diagnosed within 5 years prior to initial administration, exceptions include radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radical resection of carcinoma in situ;
13. Symptoms of central nervous metastasis
14. A history of noninfectious pneumonia requiring glucocorticoid therapy or current interstitial lung disease within 1 year prior to initial administration;
15. Active infections that require systemic treatment;
16. A known presence of mental illness or substance abuse conditions that may affect compliance with the test requirements;
17. Human immunodeficiency virus (HIV) infection；
18. Untreated active hepatitis B；
19. Active subjects with HCV infection；
20. vaccine was administered within 30 days prior to initial administration (cycle 1, day 1)；
21. Medical history or evidence of disease, abnormal values of treatment or laboratory tests, or other conditions deemed inappropriate by the Investigator to interfere with the results of the study, prevent subjects from participating fully in the study;
22. breastfeeding women. Patients with previous and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe pulmonary impairment, etc.;
23. Patients whose cardiopulmonary function cannot tolerate anesthesia；
24. The investigator evaluates other circumstances that may affect the conduct of the clinical study and the judgment of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2025-08-03 (Estimated); Study Completion 2025-08-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing clinical and laboratory adverse events (AEs) | 1 year
  Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0.
Objective Response Rate | 5 years
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study.
Measurement of CD4/CD8 T lymphocyte subsets. | 3 years
  CD4/CD8 T lymphocyte subsets were detected by flow cytometry.
The IFN-γ T cells responses induced by neoantigen | 2 years
  The response of IFN-γ T cells induced by neoantigen was detected by ELispot.

SECONDARY OUTCOMES:
Overall Survival(OS) | 5 years
  Time from surgery to death or last follow-up.
Progression-free Survival(PFS) | 3 years
  Time from surgery to any progression.
Peripheral blood T cell receptor sequencing analysis | 2 years
  The diversity and clonability of T cells were analyzed by peripheral blood T cell receptor sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Fang Y, Mo F, Shou J, Wang H, Luo K, Zhang S, Han N, Li H, Ye S, Zhou Z, Chen R, Chen L, Liu L, Wang H, Pan H, Chen S. A Pan-cancer Clinical Study of Personalized Neoantigen Vaccine Monotherapy in Treating Patients with Various Types of Advanced Solid Tumors. Clin Cancer Res. 2020 Sep 1;26(17):4511-4520. doi: 10.1158/1078-0432.CCR-19-2881. Epub 2020 May 21. PMID 32439700
- [Background] Ott PA, Hu-Lieskovan S, Chmielowski B, Govindan R, Naing A, Bhardwaj N, Margolin K, Awad MM, Hellmann MD, Lin JJ, Friedlander T, Bushway ME, Balogh KN, Sciuto TE, Kohler V, Turnbull SJ, Besada R, Curran RR, Trapp B, Scherer J, Poran A, Harjanto D, Barthelme D, Ting YS, Dong JZ, Ware Y, Huang Y, Huang Z, Wanamaker A, Cleary LD, Moles MA, Manson K, Greshock J, Khondker ZS, Fritsch E, Rooney MS, DeMario M, Gaynor RB, Srinivasan L. A Phase Ib Trial of Personalized Neoantigen Therapy Plus Anti-PD-1 in Patients with Advanced Melanoma, Non-small Cell Lung Cancer, or Bladder Cancer. Cell. 2020 Oct 15;183(2):347-362.e24. doi: 10.1016/j.cell.2020.08.053. PMID 33064988